CLINICAL TRIAL: NCT07219030
Title: A Phase 1, Randomized, Placebo-controlled Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Emraclidine Following Multiple Ascending Oral Doses in Healthy Elderly Subjects
Brief Title: A Study to Assess the Adverse Events and How Oral Emraclidine Moves Through the Body of Healthy Elderly Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M25-904
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-1231

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Emraclidine or Placebo- Group 1 (Experimental): Participants will receive oral doses of emraclidine or placebo for 10 days or 17 days
  Interventions: Drug: Emraclidine; Drug: Placebo
- Emraclidine or Placebo- Group 2 (Experimental): Participants will receive oral doses of emraclidine or placebo for 10 days or 17 days
  Interventions: Drug: Emraclidine; Drug: Placebo
- Emraclidine or Placebo- Group 3 (Experimental): Participants will receive oral doses of emraclidine or placebo for 10 days or 17 days.
  Interventions: Drug: Emraclidine; Drug: Placebo
- Emraclidine or Placebo- Group 4 (Experimental): Participants will receive oral doses of emraclidine or placebo for 10 days or 17 days.
  Interventions: Drug: Emraclidine; Drug: Placebo

INTERVENTIONS:
Drug: Emraclidine — Oral tablets
Drug: Placebo — Oral tablets

SUMMARY:
This study is to assess how oral emraclidine moves through the body of healthy elderly adult participants, and assess adverse events, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* BMI is ≥ 18.0 to ≤ 32.0 kg/m2 after rounding to the tenths decimal at Screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Body weight > 45 kg at the time of screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, genitourinary, immunological, hematologic, neurological or psychiatric disease or disorder, or any other uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.
* Evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than successfully treated non-metastatic cutaneous squamous cell, basal cell carcinoma or localized carcinoma in situ of the cervix.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to approximately 50 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Number of Participants with Clinical Significant Change From Baseline in Vital Sign Measurements | Up to approximately 20 days
  Number of participants with clinical significant change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Number of Participants with Clinical Significant Change from Baseline in Electrocardiogram (ECG) | Up to approximately 20 days
  12-lead resting ECG will be recorded.
Number of Participants with Clinical Significant Change in Physical Examinations | Up to approximately 20 days
  Number of participants with clinical significant change in physical examinations will be assessed.
Number of Participants with Clinical Significant Change in Clinical Laboratory Test Results Like Hematology will be Assessed | Up to approximately 20 days
  Number of participants with clinical significant change in clinical laboratory test results will be assessed.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately 20 days
  The C-SSRS is a clinician-rated instrument that reports the severity of both suicidal ideation and behavior, with a higher score denoting more severe suicidal ideation and behavior.
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) | Up to approximately 20 days
  AIMS assesses abnormal involuntary movements, such as tardive dyskinesia, associated with antipsychotic drugs; it measures facial, oral, extremities, and trunk movements, as well as the participant's awareness of abnormal movements. The first 10 items are rated on a none (0) to severe (4) scale. There are an additional 2 items on dental status that are answered yes or no.
Change From Baseline in Barnes Akathisia Rating Scale (BARS) | Up to approximately 20 days
  BARS is a 4-item rating scale used to assess drug-induced akathisia. The scale comprises items for rating the observable restless movements that characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia (each on a 4-point scale from normal [0] to severe [3]). In addition, there is a global severity for akathisia rated on a 6-point scale (absent [0] to severe akathisia [5]).
Change From Baseline in Simpson-Angus Scale (SAS) | Up to approximately 20 days
  SAS is a 10-item rating scale for assessment of antipsychotic-induced parkinsonism in both clinical practice and research settings. Each item ranges from 0 (normal) to 4 (extreme symptoms). The scale consists of 1 item measuring gait (hypokinesia), 6 items measuring rigidity, and 3 items measuring glabella tap, tremor, and salivation, respectively.
Maximum Observed Plasma Concentration (Cmax) of Emraclidine | Up to approximately 20 days
  Cmax of Emraclidine
Maximum Observed Plasma Concentration (Cmax) of Metabolite (CV-0000364) | Up to approximately 20 days
  Cmax of Metabolite (CV-0000364)
Time to Cmax (Tmax) of Emraclidine | Up to approximately 20 days
  Tmax of Emraclidine
Time to Cmax (Tmax) of Metabolite (CV-0000364) | Up to approximately 20 days
  Tmax of Metabolite (CV-000036)
Area Under the Concentration-Time Curve from Time 0 to Time t (AUCt) of Emraclidine | Up to approximately 20 days
  AUCt of Emraclidine
Area Under the Concentration-Time Curve from Time 0 to Time t (AUCt) Metabolite (CV-000036) | Up to approximately 20 days
  AUCt of Metabolite (CV-000036)
Area under the plasma concentration-time curve over the dosing interval (AUCtau) of Emraclidine | Up to approximately 20 days
  AUCtau of Emraclidine
Minimum plasma concentration (Cmin) of Emraclidine | Up to approximately 20 days
  Cmin of Emraclidine
Minimum plasma concentration (Cmin) of Metabolite (CV-0000364) | Up to approximately 20 days
  Cmin of Metabolite (CV-0000364)
Average plasma concentration (Cavg) of Emraclidine | Up to approximately 20 days
  Cavg of Emraclidine
Average plasma concentration (Cavg) of Metabolite (CV-0000364) | Up to approximately 20 days
  Cavg of Metabolite (CV-0000364)
Metabolite to Parent Ratio (MRCmax) of Emraclidine | Up to approximately 20 days
  MRCmax of Emraclidine calculated from Cmax
Metabolite to Parent Ratio (MRCmax) of Metabolite (CV-0000364) | Up to approximately 20 days
  MRCmax of Metabolite (CV-0000364) calculated from Cmax
Metabolite to Parent Ratio (MRAUCtau) of Emraclidine | Up to approximately 20 days
  MRAUCtau of Emraclidine based on AUCtau
Metabolite to Parent Ratio (MRAUCtau) of Metabolite (CV-000036) | Up to approximately 20 days
  MRAUCtau of Metabolite (CV-000036) based on AUCtau
Terminal Phase Elimination Half-Life (t1/2) of Emraclidine | Up to approximately 20 days
  Terminal phase elimination half-life of Emraclidine
Terminal Phase Elimination Half-Life (t1/2) of Metabolite (CV-000036) | Up to approximately 20 days
  Terminal phase elimination half-life of Metabolite (CV-000036)
Apparent terminal phase elimination constant (β) of Emraclidine | Up to approximately 20 days
  β of Emraclidine
Apparent terminal phase elimination constant (β) of Metabolite (CV-0000364) | Up to approximately 20 days
  β of Metabolite (CV-0000364)
Peak-to-trough ratio (PTR) of Emraclidine | Up to approximately 20 days
  PTR of Emraclidine
Peak-to-trough ratio (PTR) of Metabolite (CV-000036) | Up to approximately 20 days
  PTR of Metabolite (CV-000036)
Accumulation ratio for Cmax (RacCmax) of Emraclidine | Up to approximately 20 days
  RacCmax of Emraclidine
Accumulation ratio for Cmax (RacCmax) of Metabolite (CV-0000364) | Up to approximately 20 days
  RacCmax of Metabolite (CV-0000364)
Accumulation ratio for AUCtau (RacAUCtau) of Emraclidine | Up to approximately 20 days
  RacAUCtau of Emraclidine
Accumulation ratio for AUCtau (RacAUCtau) of Metabolite (CV-0000364) | Up to approximately 20 days
  RacAUCtau of Metabolite (CV-0000364)
Apparent Clearance of Drug from Plasma (CL/F) of Emraclidine | Up to approximately 20 days
  CL/F of Emraclidine
Apparent Volume of Distribution DuringTerminal Phase (Vz/F) of Emraclidine | Up to approximately 20 days
  Vz/F of Emraclidine
Area under the plasma concentration-time curve over the dosing interval (AUCtau) of Metabolite (CV-0000364) | Up to approximately 20 days
  AUCtau of Metabolite (CV-0000364)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (4):
  - Altasciences Clinical Los Angeles /ID# 276854, Cypress, California
  - K2 Medical Research, LLC /ID# 276636, Maitland, Florida
  - Clinical Pharmacology Of Miami /ID# 276856, Miami, Florida
  - Acpru /Id# 276996, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-904